CLINICAL TRIAL: NCT06524583
Title: Interest of Adjuvant Chemotherapy in Patients With CINSARC High-risk Localized Resected Uterine Leiomyosarcoma - Sarcome 15
Brief Title: Interest of Post-operative Chemotherapy in Patients With Localised Uterine Leiomyosarcoma Suspected of Having a High Risk of Recurrence Based on a Biological Test Performed on the Tumour
Acronym: L-UteCIN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: PharmaMar (Industry); Ligue contre le cancer, France (Other); National Research Agency, France (Other); University Hospital, Marseille (Other); Institut Claudius Regaud (Other); Institut Bergonié (Other); Oncopole (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UC-SAR-2212; 2023-506350-21-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Leiomyosarcoma Uterus
MeSH Terms: interventions — Doxorubicin; Trabectedin

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized and comparative phase II trial and prospective cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (No Intervention): Standard of care : Active surveillance
- Arm B (Experimental): Experimental treatment: 4 cycle of Doxorubicine + trabectedin
  Interventions: Drug: Doxorubicin; Drug: Trabectedin
- Prospective Cohort (No Intervention): Standard of care : Active surveillance

INTERVENTIONS:
Drug: Doxorubicin — 60 mg/m² intravenous (IV) at Day 1 every 3 weeks (4 cycles)
  Arms: Arm B
Drug: Trabectedin — 1.1 mg/m² intravenous (IV) at Day 1 every 3 weeks (4 cycles)
  Other Names: Yondelis
  Arms: Arm B

SUMMARY:
Addition of postoperative chemotherapy to prevent or delay recurrence in patients newly diagnosed with localized uterine leiomyosarcoma and who have undergone complete tumor surgery.

DETAILED DESCRIPTION:
This is a biological driven study comprising:

* a multicenter, randomized and comparative phase II trial designed to demonstrate whether adding 4 cycles of post-operative chemotherapy improves relapse-free survival as compared with follow-up (standard management) in patients with resected FIGO stage I uterine leiomyosarcoma, considered at high-risk according to CINSARC NanoCind® signature.
* a prospective cohort for patients with resected FIGO stage I uterine leiomyosarcoma, considered at low-risk according to CINSARC NanoCind® signature.

HIGH-RISK (HR) CINSARC patients will be randomized post-operatively between the two arms of treatment, i.e. standard treatment (active post-surgical surveillance) or chemotherapy, with a 1:1 randomization on one factor: morcellation versus no morcellation of uterine tumor.

LOW-RISK (LR) CINSARC patients' data will be prospectively collected

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have a histologically confirmed diagnosis of uterine leiomyosarcoma obtained less than 8 weeks from the surgery
2. Eastern cooperative oncology group (ECOG) performance status (PS) 0 or 1
3. Patient was previously untreated with chemotherapy for a sarcoma, and did not receive anthracyclines and/or trabectedin for another cancer
4. Available Formalin Fixed Paraffin Embedded (FFPE) tumor blocks in sufficient quantity and quality to allow CINSARC NanoCind® qualification (low-risk or high-risk)
5. Age ≥ 18 years and ≤ 75 years
6. FIGO 2018 classification stage I (IA and IB), with complete resection (total hysterectomy and optional bilateral oophorectomy; possible ovarian preservation is feasible in selected cases)
7. No measurable disease, as assessed by the investigator: normal post-operative thoracic, abdominal and pelvic CT-scan or normal MRI of abdomen and pelvis + normal chest CT performed within 4 weeks prior to inclusion or randomization in the study
8. Signed informed consent form prior to any trial specific procedures consistent with international conference on harmonisation - good clinical practice (ICH-GCP) and local legislation
9. Patient must be affiliated to a social security system or in possession of equivalent private health insurance (according to local regulations for participation in clinical trials).

   Additional inclusion criteria for randomization
10. Inclusion criteria checked at study entry are all still met at the time of randomization
11. High-risk CINSARC signature
12. Patient must have a diagnosis of uterine leiomyosarcoma confirmed by a local sarcoma expert pathologist from RRePS (Sarcoma Pathology Reference Network from NETSARC +) locally or by the study central RRePS expert pathologist.
13. Adequate hematologic organ function:

    * absolute neutrophil count ≥ 1.5 Giga/ L
    * hemoglobin ≥ 9 g/dL
    * platelets ≥ 100 Giga/L
14. Adequate renal function: serum creatinine ≤ 1.5 mg/dL (≤ 132.6 µmol/L) or calculated creatinine clearance ≥60 mL/min (by the Cockcroft and Gault formula)
15. Adequate liver function: total bilirubin ≤ upper limit of normal (ULN), transaminases ≤ 2.5 x ULN, alkaline phosphatases ≤ 1.5 x ULN
16. Adequate cardiac function: cardiac ultrasound and/or isotopic ventriculography, shortening fraction (SF) > 30%, Left Ventricular Ejection Fraction (LVEF) (per ultrasound or scintigraphy) > 50%
17. Creatine phosphokinase (CPK) ≤ 2,5 x ULN
18. Albumin ≥ 25 g/L
19. Signed informed consent form for the randomized phase, consistent with ICH-GCP and local legislation.

Exclusion Criteria:

* Exclusion criteria:

  1. All other histology types of uterine sarcoma (adenosarcoma, endometrial sarcoma, undifferentiated uterine sarcoma)
  2. Prior or concurrent malignant disease diagnosed or treated in the last 5 years except for adequately treated in situ carcinoma of the cervix, basal or squamous skin cell carcinoma, or in situ transitional bladder cell carcinoma
  3. Planned pelvic post-operative radiation therapy
  4. Metastatic or measurable disease on CT-Scan
  5. Known hypersensitivity to doxorubicin or trabectedin or to any of the excipients
  6. Any contra-indication for the use of doxorubicin and/or trabectedin treatment
  7. Participation in another therapeutic trial within the 30 days prior to inclusion in the study
  8. Active viral hepatitis B or C or known human immunodeficiency virus (HIV) infection.
  9. Prior anticancer therapy, including radiotherapy, endocrine therapy, immunotherapy, chemotherapy (CT) or other investigational agents within the last 4 weeks (6 weeks for nitrosoureas and mitomycin C)
  10. Cardiovascular dysfunction:
* Congestive heart failure (New York Heart Association [NYHA]) ≥ 2)
* Myocardial infarction <6 months before study
* Poorly controlled cardiac arrhythmias
* Uncontrolled hypertension
* Unstable (angina symptoms at rest) or new-onset angina (begun within the last 3 months) 11. Ongoing infection > Grade 2 according to NCI-CTCAE v5.0 12. Breastfeeding woman 13. Patients unwilling or unable to comply with the medical procedures and follow-up required by the trial because of geographic, familial, social, or psychological reasons 14. Persons deprived of their liberty or under protective custody or guardianship.

Additional exclusion criteria for randomization 15. At least one of the exclusion criteria check at study entry is met at the time of randomization 16. Unknown risk for CINSARC signature 17. For patients who require a pathological review by the study central pathologist, failure to obtain a confirmed diagnosis at randomization 18. More than 13 weeks have elapsed since the surgery procedure. 19. Patient receiving phenytoin within 88 hours prior to randomisation and or live attenuated vaccines within 14 days prior to randomisation and or CYP3A4 inhibitors (e.g. oral ketoconazole, fluconazole, ritonavir, clarithromycin or aprepitant) and or strong CYP3A4 inducers (e.g. rifampicin, phenobarbital, St John's wort).

Criteria for continuing in the prospective cohort :

1. Patient must have a diagnosis of uterine leiomyosarcoma confirmed by a sarcoma expert pathologist or by the study central pathologist
2. Patients with a low-risk CINSARC signature

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival | From randomization or enrollment to disease recurrence or death, up to 5 years
  The relapse-free survival is defined as the time from the date of randomization assignment (or the date of enrollment for patients in the prospective cohort) to the date of first disease recurrence/relapse (local/regional recurrence and/or distant metastasis) or death from any cause whichever comes first.

SECONDARY OUTCOMES:
Overall survival | From randomization or enrollment to death, up to 5 years
  The overall survival is the length of time from randomization (or enrollment for patients in the prospective cohort) that patients enrolled in the study are still alive.
Metastases-free survival | From randomization or enrollment to metastases onset or death, up to 5 years
  The metastases-free survival is the length of time during and after the treatment for cancer that a patient is still alive and the cancer has not spread to other parts of the body.
Incidence of adverse events | Throughout study completion, up to 5 years
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.
  Safety and tolerability (NCI-CTCAE v5.0) will be assessed through the incidence of adverse events, treatment-related adverse events, serious adverse events (SAEs); and death.
Quality of life questionnaire - Core 30 (QLQ-C30) | At baseline, end of treatment (up to week 12), 4 months, 6 months, 1 year and 2 years
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.

CONTACTS AND LOCATIONS:
Overall Officials: Florence DUFFAUD, MD, Principal Investigator — La TIMONE University Hospital
Locations (25):
- France (25):
  - Institut de Cancerologie de L'Ouest (Ico), Angers
  - Hopital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges Francois Leclerc, Dijon
  - Chu Limoges, Limoges
  - Centre Léon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - La Timone University Hospital, Marseille
  - Centre Antoine Lacassagne, Nice
  - Hopital Saint Louis, Paris
  - Hôpital Cochin, Paris
  - Groupe Hospitalier Diaconesses Croix St Simon, Paris
  - Hopital Tenon, Paris
  - Institut Curie, Paris
  - Chu de Poitiers, Poitiers
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut de cancerologie de l'ouest site Rene Gauducheau, Saint-Herblain
  - Institut de Cancerologie Strasbourg Europe (Icans), Strasbourg
  - Institut Claudius Regaud, Toulouse
  - CHU Bretonneau, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.